CLINICAL TRIAL: NCT05096962
Title: SARS-CoV-2-CZ-PREVAL-II Study
Brief Title: COVID-19: SARS-CoV-2-CZ-PREVAL-II Study
Status: Completed | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Ministry of Health, Czech Republic (Other Government); The National Institute of Public Health (Unknown); The Institute of Molecular and Translational Medicine, Czech Republic (Other); University Hospital Olomouc (Other); Institute for Clinical and Experimental Medicine (Other Government); Thomayer University Hospital (Other); Czech Academy of Sciences (Other); Palacky University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/2
Record Dates: First submitted 2021-10-22; First posted 2021-10-27 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: antibodies; cell immunity
MeSH Terms: conditions — COVID-19 | interventions — Immunity, Cellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma sampling will be archived in the biobank for subsequent analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm IKEM: Arm IKEM (Institute for Clinical and Experimental Medicine) is represented by two subcohorts:
  * participants with chronic illness (adults only), which are part of the research project of the Institute of Clinical and Experimental Medicine (the expected number of participants in the study - 3 000)
  * healthy subjects from the Study of Czech Academy of Science, who are following up in the Institute of Clinical and Experimental Medicine (the expected number of subjects in the study - 2000) The subjects will be contacted based on the Hospital study database.
  Interventions: Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies; Diagnostic Test: Cellular immunity
- Arm FTN: Arm FTN (Thomayer University Hospital) is represented by the healthcare staff of the Hospital (the expected number of subjects in the study - 1800).
  Interventions: Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies; Diagnostic Test: Cellular immunity
- Arm Olomouc: Arm Olomouc is represented by participants, who participated in the Study "Herd Immunity Study SARS-CoV-2-CZ-Preval" in May 2020 and at the same time subjects who will be willing to participate in this study. The involvement of subjects from two localities is expected:
  * Olomouc
  * Litovel, Uničov and Červenka. The expected number of subjects in the study is approximately 2500.
  Interventions: Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies; Diagnostic Test: Cellular immunity

INTERVENTIONS:
Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies — The study will evaluate the current presence of infection, specific antibodies at least in the IgG class in blood plasma or serum (antibody tests focusing on two SARS-CoV-2 proteins: S-protein and N-protein).
Diagnostic Test: Cellular immunity — Quantification of the level of cellular immunity from venous blood collected in approximately 30% of examined individuals.

SUMMARY:
The aim of the SARS-CoV-2-CZ-PREVAL-II Study is to quantify the prevalence of participants with antibodies against SARS-CoV-2 and/or cell immunity against SARS-CoV-2 in specific subjects cohorts.

DETAILED DESCRIPTION:
The aim of the SARS-CoV-2-CZ-PREVAL-II Study is to quantify the prevalence of participants with antibodies against SARS-CoV-2 and/or cell immunity against SARS-CoV-2 in four specific cohorts: participants with chronic illness, healthy volunteers participating in the Study of the Czech Academy of Science, healthcare workers, and healthy volunteers that participated in the "Herd Immunity Study SARS-CoV-2-CZ-Preval" in May 2020.

The primary aim of the study is to estimate the number of people with anti-SARS-CoV-2-antibodies, i.e., people with COVID-19 history, or with vaccination against COVID-19.

Antibodies test will focus on two main proteins of virus SARS-CoV-2: S-protein and N-protein.

The secondary aims of the study are:

* quantitative analysis of cellular immunity and the other relevant markers,
* estimation of the proportion of participants with asymptomatic COVID-19 infection
* quantification of anti-SARS-CoV-2 antibodies and cell immunity according to individual risk factors.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed consent
* willingness to complete the study questionnaire
* demographic criteria - age 18 years old and more
* clinical criteria - without acute health problems
* time criteria - sample collection in the defined period time

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of different cohorts of people. The first cohort, Arm IKEM, is chosen from a database of chronically ill patients and subjects involved in the sociological study of the Czech Academy of Sciences. The second cohort, Arm FTN, is chosen from healthcare workers of the Thomayer University Hospital. The third cohort, Arm Olomouc, is composed of volunteers who participated in the Study SARS-CoV-2-CZ-Preval in May 2020.
  All subjects will be contacted by email, phone, or SMS.
Sampling Method: Non-Probability Sample
Enrollment: 7268 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Detection of a number of subjects with IgG anti-SARS-CoV-2 antibodies | September-October 2021
  The primary outcome is to quantify the prevalence of participants with IgG anti-SARS-CoV-2 antibodies in the specified subjects cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Marián Hajdúch, Assoc. Prof., Principal Investigator — Institute of Molecular nad Translational Medicine; Věra Adámková, Prof., Principal Investigator — Institute for Clinical and Experimental Medicine; Markéta Ibrahimová, Ph.D., Principal Investigator — Thomayer University Hospital; Barbora Macková, M.D., Principal Investigator — The National Institute of Public Health; Ladislav Dušek, Prof., Study Director — Institute of Health Information and Statistics of the Czech Republic
Locations (1):
- Institute of Health Information and Statistics of the Czech Republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.